CLINICAL TRIAL: NCT00386711
Title: A Study on Improving Detection and Management of Suicide Risk Among Depressed Patients in Primary Care
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NBH038
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-10

CONDITIONS: Depression; Suicide
Keywords: suicide; depressed patients; primary care
MeSH Terms: conditions — Depression; Suicide

INTERVENTIONS:
Behavioral: training on identification of suicide risk and depression

SUMMARY:
improve detection and management of suicide risk among depressed patients in primary care

DETAILED DESCRIPTION:
After intervention of training on the identification and management of depression and suicide risk in primary health care professionals, the ability of detection and management of suicide risk among depressed patients in primary care is expected to be improved compared to baseline evaluation.

ELIGIBILITY:
Inclusion Criteria:

* consecutive outpatient

Exclusion Criteria:

* severe physical conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2160
Dates: Start 2006-10; Study Completion 2007-01

PRIMARY OUTCOMES:
Kappa of diagnostic consistency

SECONDARY OUTCOMES:
ratio of optimal managment

CONTACTS AND LOCATIONS:
Overall Officials: SHUTAO ZHAI, DOCTOR, Study Director — Nanjing Brain Hospital
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China